CLINICAL TRIAL: NCT02166177
Title: Pilot Study Evaluating the Safety and Efficacy Profile of Regulatory T Cell Therapy in Liver Transplant Recipients
Brief Title: Safety and Efficacy Study of Regulatory T Cell Therapy in Liver Transplant Patients
Acronym: ThRIL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Treg Liver Trial
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: End-stage Liver Disease
MeSH Terms: conditions — End Stage Liver Disease

ARMS (1):
- Autologous Regulatory T cell therapy (Experimental): Autologous regulatory T cell therapy infused intravenously (2 dose groups: low dose and high dose)
  Interventions: Drug: Autologous regulatory T cell product

INTERVENTIONS:
Drug: Autologous regulatory T cell product — Autologous regulatory T cell therapy infused intravenously (2 dose groups: low dose and high dose). The patients also receive rabbit Antithymocyte Globulin (rATG), tacrolimus, and sirolimus.

SUMMARY:
'ThRIL' aims to explore the feasibility, safety and efficacy of TR002, a regulatory cell therapy, as adjunct immunosuppressive treatment in the context of liver transplantation

DETAILED DESCRIPTION:
Stage I: To evaluate the safety of administering TR002 to liver transplant recipients.

Stage II: To evaluate the efficacy of TR002 administration in allowing for the discontinuation of immunosuppressive therapy in liver transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* adult patients with end-stage liver disease listed for primary liver transplant;
* calculated MELD score ≤ 25 at time of transplantation

Exclusion Criteria:

* HIV or RNA-positive Hepatitis C Virus infection;
* autoimmune liver disease
* previous organ transplant
* Ebstein Virus and/or Cytomegalovirus sero-negativity
* chronic use of systemic immunosuppressants
* hepatocellular carcinoma outside Milano criteria
* leukocytes <1.5x10^9/L and/or platelets <50x10^9/L.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-06; Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities (DLTs) | 1 month after IMP administration
  rate of adverse events qualifying as dose limiting toxicities
Graft Loss | 24 months
  Rate of cellular rejection

SECONDARY OUTCOMES:
Immunosuppressive doses | 24 months
  total dose of immunosuppressive medication administered
Prevention of acute and chronic rejection | 24 months
  incidence of rejection episodes
Acute and Chronic Toxicity | 24 months
  incidence of immunological reactions, biochemical disturbances
Liver histology | 12 months
  liver biopsy analysis
Rate of successful immunosuppressive drug withdrawal | 24 months
  total dose of immunosuppressive medication administered

OTHER OUTCOMES:
Immunological biomarkers | 12 months
  immune monitoring analysis of blood samples investigating the effect of TR002 on blood cell immunophenotype

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Lombardi, PhD, Study Director — King's College London
Locations (1):
- Kings College Hospital, London, United Kingdom